CLINICAL TRIAL: NCT00106067
Title: Aging and Family Outcomes in Supportive Care of Advanced Cancer Patients
Acronym: A&SC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIR 03-255
Record Dates: First submitted 2005-03-18; First posted 2005-03-21 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Aging; Neoplasms
Keywords: aging; behavioral research; quality of life; end of life; family relations; supportive care; advanced care; bereavement
MeSH Terms: conditions — Neoplasms; Death | interventions — Coping Skills; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): In the intervention arm, Patients and their family caregivers have access to a coping and communication support practitioner (CCSP) (see intervention description) in addition to receiving the usual care in the site.
  Interventions: Behavioral: coping and communication support (CCS) intervention
- Arm 2 (No Intervention): In the control arm, Patients are receiving the usual care in the site.

INTERVENTIONS:
Behavioral: coping and communication support (CCS) intervention — Trained clinical nurse specialists with masters� degrees in mental health will serve as CCS practitioners and they will be available to patients and family caregivers on a 24/7 basis to assist with coping and communication challenges as they may arise.
  The CCS intervention is tailored to individual preferences over time, and designed to accommodate different age groups, especially older adults and their families.
  Arms: Arm 1

SUMMARY:
The diagnosis of advanced, incurable cancer at different stages of the adult life span holds a variety of meanings for family members who often must play critical roles in patient care and decision-making. Family caregivers are greatly affected by the diagnosis and treatment of late-stage cancer in a loved one and may find it difficult to meet the demands of taking care of their loved one through end-of-life care and taking care of their own well-being. This grant provides funding to examine processes and outcomes of the intervention for family caregivers of advanced cancer patients.

DETAILED DESCRIPTION:
We are testing a coping and communication support (CCS) intervention for advanced stage cancer patients and their family caregivers over the period when goals of care may shift, i.e. beginning shortly after diagnosis. This randomized clinical trial is being conducted in two urban tertiary cancer clinics that reach patients and families in low income and diverse underserved populations: the Louis Stokes Cleveland VAMC and MetroHealth Medical Center. Recruitment and randomization are based on patient's diagnosis and age. The patient had to have been diagnosed with a stage IV cancer within a year of enrollment and they must fall into one of two age groups: middle-aged (ages 40-60); or older (61 and older). Patients are stratified by age group and then randomized to usual care or CCS intervention. Family care-givers are randomized along with the patient. Trained clinical nurse specialists with advanced training in mental health serve as CCS practitioners. They are available to patients and family caregivers on a 24/7 basis to assist with coping and communication challenges as they may arise. The primary goal of this project is to examine main effects of the intervention and patient age group interaction effects of the CCS intervention on perspectives and well-being of family caregivers during advanced cancer care and in bereavement.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed within 1 year with advanced cancer (stage IV), aged 40 years or older.
* Patients must be cognitively intact at time of enrollment.
* Patient need not have family care-giver to be enrolled, but if there is one, FCG is enrolled with the patient. FCG need not be 40 years of age.

Exclusion Criteria:

- Less than stage IV cancer, stage IV cancer diagnosed over 1 year previously or younger than 40 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2004-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The primary goal of this project is to examine main effects of the intervention and patient age group interaction effects of the CCS intervention on perspectives and well-being of family caregivers during advanced cancer care and in bereavement. | one year

SECONDARY OUTCOMES:
To assess the efficacy of the intervention among patients in coping and decisions around end of life. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Julia Rose, PhD MA, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

REFERENCES:
- [Result] Bowman KF, Rose JH, Radziewicz RM, O'Toole EE, Berila RA. Family caregiver engagement in a coping and communication support intervention tailored to advanced cancer patients and families. Cancer Nurs. 2009 Jan-Feb;32(1):73-81. doi: 10.1097/01.NCC.0000343367.98623.83. PMID 19104204
- [Result] Rose JH, Radziewicz R, Bowmans KF, O'Toole EE. A coping and communication support intervention tailored to older patients diagnosed with late-stage cancer. Clin Interv Aging. 2008;3(1):77-95. doi: 10.2147/cia.s1262. PMID 18488881
- [Result] Rose JH, O'Toole EE, Einstadter D, Love TE, Shenko CA, Dawson NV. Patient age, well-being, perspectives, and care practices in the early treatment phase for late-stage cancer. J Gerontol A Biol Sci Med Sci. 2008 Sep;63(9):960-8. doi: 10.1093/gerona/63.9.960. PMID 18840801